CLINICAL TRIAL: NCT06241144
Title: Information and Communication Technology -Based Health Behavior Change Support System to Modify Lifestyle After Delivery: Randomized Controlled Intervention Study
Brief Title: Supporting Lifestyle Changes After Delivery
Acronym: STELLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Principal Investigator, Marja Vääräsmäki, Professor, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39/2023
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Maternal; Lifestyle
MeSH Terms: conditions — Pregnancy in Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Information and communication technology -based health behavior change support system
- Control (No Intervention)

INTERVENTIONS:
Device: Information and communication technology -based health behavior change support system — Information and communication technology -based health behavior change support system addition to conventional postpartum lifestyle education
  Arms: Intervention

SUMMARY:
Use of information and communication technology -based health behavior change support system in modifying lifestyle after delivery among women with obesity.

DETAILED DESCRIPTION:
Postpartum weight retention is common and particular when accompanied with prior obesity, it further increases the risks of subsequent pregnancies and adverse effects on the long-term health.

The aim of this randomized controlled trial is to examine whether using an information and communication technology (ICT) -based health behavior change support system (HBCSS) reduce postpartum weight retention and disorders related to subsequent pregnancy. Web-based HBCSS application utilizes persuasive design and cognitive behavioral therapy.

200 participants with prepregnancy obesity (BMI ≥ 30.0 kg/m^2) and age ≥ 18 years are randomly assigned into two groups after delivery in the Oulu university hospital. The study period begins 5-12 weeks after delivery. All participants will have conventional postpartum lifestyle counselling and the intervention group get in addition access for 12 months to web-based HBCSS application, which is recommended to use twice a week for 5-10 minutes.

Participants are followed by questionnaires up to 24 months. The main outcome is weight change from baseline to 12 and 24 months. Medical records and national registers are used for long-term follow-up. Researchers have permission to contact participants afterwards. The ethical approval is permitted by the Regional Medical Research Ethics Committee of the Wellbeing Services County of North Ostrobothnia. The authorization for the use of medical device is granted from the Finnish Medicines Agency. Recruitment of the participants will be performed 2/2024-1/2026.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy BMI ≥ 30.0 kg/m^2
* Smartphone user

Exclusion Criteria:

* Eating disorder
* Severe mental disorder
* Use of other lifestyle support system or medication
* Non-Finnish speaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | 12 months
  Weight change in kilograms and change of body mass index (kg/m^2)
Weight change | 24 months
  Weight change in kilograms and change of body mass index (kg/m^2)

SECONDARY OUTCOMES:
Weight change before subsequent pregnancy | 1-8 years
  Weight change in kilograms and change of body mass index (kg/m^2)
Pregnancy disorders in subsequent pregnancy (gestational diabetes, pre-eclampsia, gestational hypertension, preterm delivery) | 1-8 years
  Number of participants with pregnancy disorders in subsequent pregnancy (gestational diabetes, pre-eclampsia, gestational hypertension, preterm delivery, mortality)
Neonatal outcome in subsequent pregnancy (preterm birth, large for gestational age, small for gestational age, need for neonatal intensive care, mortality) | 1-8 years
  Number of neonates with adverse neonatal outcome (preterm birth, large for gestational age, small for gestational age, need for neonatal intensive care, mortality)

CONTACTS AND LOCATIONS:
Overall Officials: Marja Vääräsmäki, Professor, Principal Investigator — Research Unit of Clinical Medicine, University of Oulu, Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: STELLA project page — https://www.oulu.fi/fi/node/37815